CLINICAL TRIAL: NCT03169530
Title: Moderate Alcohol and Cardiovascular Health Trial
Acronym: MACH15
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: NIH decision
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Harvard School of Public Health (HSPH) (Other); Wake Forest University Health Sciences (Other); Julius Center (Other)
Responsible Party: Principal Investigator, Kenneth Mukamal, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017P000333; U10AA025286 (NIH)
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Results first posted 2019-01-30 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Cardiovascular Diseases; Diabetes
Keywords: cardiovascular, alcohol, diabetes
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus | interventions — Ethanol; Beer; Wine

STUDY DESIGN:
Intervention Model Description: Balanced-design randomized trial, comparing the effects of one standard serving (~15 grams) of alcohol intake daily to abstention.
Who Masked: Outcomes Assessor
Masking Description: Clinical outcome events will be assessed through medical record review by a masked Medical Safety Officer (MSO).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcohol (Active Comparator): One standard serving of alcohol (~15 gm) daily
  Interventions: Other: Alcohol
- Abstention (No Intervention): Abstention from alcohol

INTERVENTIONS:
Other: Alcohol — ~15 gm daily of beer, wine, or spirits for ~6 years
  Other Names: ethanol, beer, wine, spirits
  Arms: Alcohol

SUMMARY:
The Moderate Alcohol and Cardiovascular Health Trial (MACH15) is a multicenter, worldwide, randomized clinical trial of ~15 gm of alcohol daily versus abstention, using a balanced parallel design and single-blind assessment of all outcomes among approximately 7,800 participants aged 50 years and older with advanced cardiovascular risk. Intervention will average 6 years in duration with a common close-out date. Following recruitment and pre-screening, participants will attend a screening visit followed by a two-week abstention washout period, a baseline visit and randomization, and subsequent visits at 3 months, 6 months, 12 months, and then annually until close-out.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥50 years at screening
* Postmenopausal, defined as 12 consecutive months without menstruation
* Not alcohol naïve, defined by having consumed at least one drink of alcohol in the past five years
* High risk for the occurrence of a new cardiovascular disease event, defined as having any one of the following:

  1. American Heart Association (AHA)/American College of Cardiology (ACC) Risk Score ≥15% within the past 24 months (among those without clinical or subclinical cardiovascular disease [CVD])
  2. Clinical CVD (more than 6 months prior to randomization), defined by:

     1. Previous myocardial infarction (MI), percutaneous coronary intervention (PCI), coronary artery bypass grafting (CABG), carotid endarterectomy (CE), carotid stenting;
     2. Peripheral artery disease (PAD) with revascularization;
     3. Acute coronary syndrome with or without resting electrocardiogram (ECG) change, ECG changes on a graded exercise test (GXT), or positive cardiac imaging study;
     4. Prior stroke documented on brain imaging or with a persistent deficit.
  3. Subclinical CVD, confirmed in available medical records:

     1. At least a 50% diameter stenosis of a coronary, carotid, or lower extremity artery;
     2. Coronary artery calcium score ≥400 Agatston units;
     3. Ankle brachial index (ABI) ≤0.90;
     4. Left ventricular hypertrophy (LVH) by ECG (based on computer reading), echocardiogram report, or other cardiac imaging procedure report;
     5. Abdominal aortic aneurysm (AAA) ≥5 cm with or without repair.

Exclusion Criteria:

* High alcohol consumption, defined by any one of the following:

  1. Alcohol Use Disorders Identification Test (AUDIT) score >5 at screening
  2. Drinking, on average, >7 alcoholic beverages/week during the past 6 months
  3. Drinking 6 or more alcoholic beverages on one occasion during the past 6 months
* Yale-Brown Obsessive Compulsive Scale-heavy drinking (Y-BOCS-hd) total score of ≥6 on questions 7, 8, and 10
* Cardiovascular disease event (MI, revascularization procedure, or stroke) within the 6 months prior to randomization
* AHA Class III-IV heart failure
* History of alcohol or substance abuse (medical record confirmed or self-reported history)
* Other intolerance or allergy to alcohol
* Dual antiplatelet therapy
* History of gastric bypass surgery
* Any serious chronic liver disease (e.g., active hepatitis B and C infections) or liver tests (aspartate aminotransferase [AST], alanine aminotransferase [ALT] and gamma-glutamyl transpeptidase [GGT]) >2 times the upper limit of the normal range using local standards
* Personal history of any colon or liver cancer
* Any other cancer with a life expectancy of less than 3 years
* Diagnosed with breast cancer that required either surgery or removal of breast tissue or chemotherapy
* Mother or sister ever diagnosed with breast cancer that required either surgery or removal of breast tissue or chemotherapy
* Estimated glomerular filtration rate (eGFR) <30 ml/min /1.73m2 or end-stage renal disease (ESRD)
* Ongoing use of any medication for which alcohol consumption is contraindicated
* A Patient Health Questionnaire (PHQ-9) ≥15 at screening
* History of any organ transplant
* Unintentional weight loss >10% in last 6 months
* Currently participating in another clinical trial (intervention trial) with CVD outcomes. Note: Participant must wait until the completion of his/her activities or the completion of the other trial before being screened for MACH15. Local restrictions for entry by participants can be more conservative if mandated.
* Not willing or able to provide a name and contact information for at least one additional contact person other than self
* Investigator discretion regarding appropriateness of participation or concern about intervention adherence, including:

  1. moderate - severe psychiatric illness
  2. behavioral concerns regarding likelihood of low adherence to trial protocol
  3. a medical condition likely to limit survival to less than 3 years
  4. advanced chronic disease, such as dementia, that requires 24-hour care
* Not willing or able to provide a signed and dated informed consent form
* Not willing or able to comply with all trial procedures.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J Mukamal, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (4):
- United States (2):
  - Johns Hopkins ProHealth Clinical Research Center, Baltimore, Maryland
  - Wake Forest Sticht Center on Aging, Winston-Salem, North Carolina
- Julius Clinical, Zeist, Netherlands
- Center for Bioethics and Research, Ibadan, Nigeria

IPD SHARING:
Plan to Share IPD: No
Sponsor prohibits data sharing.

REFERENCES:
- [Background] Mukamal KJ, Clowry CM, Murray MM, Hendriks HF, Rimm EB, Sink KM, Adebamowo CA, Dragsted LO, Lapinski PS, Lazo M, Krystal JH. Moderate Alcohol Consumption and Chronic Disease: The Case for a Long-Term Trial. Alcohol Clin Exp Res. 2016 Nov;40(11):2283-2291. doi: 10.1111/acer.13231. Epub 2016 Sep 30. PMID 27688006

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 103 subjects provided signed consent, 32 subjects were randomized. The additional 71 subjects were in the screening or in the run-in stage of the trial at the time of study cessation.
Pre-assignment Details: 103 subjects provided signed consent, 32 subjects were randomized. The additional 71 subjects were in the screening or run-in stages of the trial at the time of study cessation.
Period: Overall Study
Arm/Group | Alcohol | Abstention
Started | 15 | 17
Completed | 0 | 0
Not Completed | 15 | 17
Not completed — Study ended by NIH | 15 | 17

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Alcohol | Abstention | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 7 | 8
  >=65 years | 14 | 10 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] — All Randomized Participants
  Years | 73.5 (8.7) | 68.5 (10.3) | 70.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 8 | 10 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 17 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 10 | 16
  White | 8 | 7 | 15
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 0 | 1 | 1
  United States | 11 | 11 | 22
  Nigeria | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Cardiovascular Disease or Death
Description: Time from baseline to a composite endpoint comprised of the first occurrence of a non-fatal myocardial infarction, non-fatal ischemic stroke, hospitalization for angina, coronary/carotid revascularization, or all-cause mortality.
Time Frame: Every 3 months for up to 90 months or close out, or until date of death
Population: The trial was closed prior to any subject competing a 3-month visit, precluding assessment of the primary outcome. Therefore, no data for the CV disease outcome were collected or analyzed prior to study termination. No subjects died during the trial.
Arm/Group | Alcohol | Abstention
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Cardiovascular Disease
Description: Time from baseline to a composite endpoint comprised of the first occurrence of a non-fatal myocardial infarction, non-fatal ischemic stroke, hospitalization for angina, coronary/carotid revascularization, or cardiovascular mortality.
Time Frame: Every 3 months for up to 90 months or close out, or until date of death
Population: The trial was closed prior to any subject competing a 3-month visit, precluding assessment of this secondary outcome. Therefore, no data for this outcome were collected or analyzed prior to study termination. No subjects died during the trial.
Arm/Group | Alcohol | Abstention
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Diabetes
Description: Progression among normoglycemic and pre-diabetes individuals to American Diabetes Association (ADA)-defined diabetes.
Time Frame: Every 12 months for 90 months or close out, or until date of first documented occurence
Population: The trial was closed prior to any subject competing a 12-month visit, precluding assessment of this outcome. Therefore, no data for the diabetes outcome were collected or analyzed prior to study termination.
Arm/Group | Alcohol | Abstention
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Hard Cardiovascular Disease or Death
Description: Time from baseline to a composite endpoint comprised of the first occurrence of a non-fatal myocardial infarction, non-fatal ischemic stroke, or cardiovascular death.
Time Frame: Every 3 months for 90 month or close out, or until date of death
Population: The trial was closed prior to any subject competing a 3-month visit, precluding assessment of this outcome. Therefore, no data for this outcome were collected or analyzed prior to study termination. No subjects died during the trial.
Arm/Group | Alcohol | Abstention
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Components of Primary Composite Endpoint
Description: Time from baseline to the first occurrence of each of the components of primary outcome (5 outcomes).
Time Frame: Every 3 months for up to 90 months or close out, or until date of death
Population: The trial was closed prior to any subject competing a 3-month visit, precluding assessment of these outcomes. Therefore, no data were collected or analyzed prior to study termination. No subjects died during the trial.
Arm/Group | Alcohol | Abstention
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Cardiovascular Death
Description: Time from baseline to cardiovascular mortality.
Time Frame: Every 3 months for 90 months or closeout, or date of death
Population: The trial was closed prior to any subject competing a 3-month visit, precluding assessment of this outcome. Therefore, no data for this outcome were collected or analyzed prior to study termination. No subjects died prior to completion of a 3-month visit.
Arm/Group | Alcohol | Abstention
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Pre-Diabetes
Description: Progression among normoglycemic individuals to ADA-defined pre-diabetes.
Time Frame: Every 12 months for 90 months or closeout
Population: The trial was closed prior to any subject competing a 12-month visit, precluding assessment of this outcome. Therefore, no data for this outcome were collected or analyzed prior to study termination.
Arm/Group | Alcohol | Abstention
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 months; from first enrolled subject until study termination.
Arm/Group | Alcohol | Abstention
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17
Other Adverse Events (participants affected / at risk) | 0/15 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT03169530/Prot_SAP_004.pdf
  • Informed Consent Form (2018-04-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT03169530/ICF_005.pdf